CLINICAL TRIAL: NCT02223000
Title: Relative Bioavailability and Tolerability of Various Experimental Formulations of 50 mg BIBV 308 SE Administered Orally Twice a Day Over 3.5 Days to Healthy Subjects (Intraindividual Comparison, Open, Partially Randomised).
Brief Title: Relative Bioavailability and Tolerability of Various Experimental Formulations of BIBV 308 SE in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 528.22
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (3):
- BIBV 308 SE solution (Active Comparator)
  Interventions: Drug: BIBV 308 SE solution
- BIBV 308 SE capsule 1 (Experimental)
  Interventions: Drug: BIBV 308 SE capsule 1
- BIBV 308 SE capsule 2 (Experimental)
  Interventions: Drug: BIBV 308 SE capsule 2

INTERVENTIONS:
Drug: BIBV 308 SE solution
  Arms: BIBV 308 SE solution
Drug: BIBV 308 SE capsule 1
  Arms: BIBV 308 SE capsule 1
Drug: BIBV 308 SE capsule 2
  Arms: BIBV 308 SE capsule 2

SUMMARY:
Comparative pharmacokinetics of 2-4 experimental modified release formulations and oral solution of BIBV 308 SE following multiple doses, tolerability

ELIGIBILITY:
Inclusion Criteria:

* Subjects that were previously entered in at least one BIBV 308 SE study to ensure that it is known how these subjects absorb BIBV 308 SE
* Healthy subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >= 18 and <= 55 years
* Broca >= -20% and <= +20 %

Exclusion Criteria:

* Poor individual absorption kinetics of BIBV 308 SE in previous studies
* Any findings of the medical examination (including blood pressure, pulse rate and Electrocardiogram (ECG)) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastro-intestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* Hypersensitivity to BIBV 308 SE and any of the excipients
* Intake of drugs with a long half-life (> 24 hours) <= 1 month prior to administration or during the trial
* Use of any drugs which might influence the results of the trial <= 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug <= 2 months days prior to administration or during the trial
* Smoker (>= 10 cigarettes or >= 3 cigars or >= 3 pipes/day)
* Inability to refrain from smoking on study days
* Known alcohol or drug abuse
* Blood donation <= 1 month prior to administration
* Excessive physical activities <= 5 days prior to administration
* History of hemorrhagic diathesis
* History of gastro-intestinal ulcer, perforation or bleeding
* History of bronchial asthma
* Any laboratory value outside the reference range of clinical relevance

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 1998-03; Primary Completion 1998-07 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma at steady state (AUCss) | up to 84 hours after drug administration
Maximum measured concentration of the analyte in plasma at steady state (Cmax,ss) | up to 84 hours after drug administration
Minimum measured concentration of the analyte in plasma at steady state (Cmin,ss) | up to 84 hours after drug administration

SECONDARY OUTCOMES:
Percent peak-trough fluctuation (%PTF) | up to 84 hours after drug administration
Time from dosing to the maximum concentration of the analyte in plasma at steady state (tmax,ss) | up to 84 hours after drug administration
Mean residence time of the analyte in the body (MRTtot) | up to 84 hours after drug administration
Apparent clearance of the analyte in plasma (CL/f) | up to 84 hours after drug administration
Ratio of Cmax,ss/AUCss | up to 84 hours after drug administration
Trough concentrations of BIBV 308 SE before doses | up to day 4